CLINICAL TRIAL: NCT00033514
Title: Phase I/II Study Of Herceptin Combined With OSI-774 In The First-Line Treatment Of Metastatic Breast Cancer Associated With HER2/Neu Overexpression
Brief Title: Trastuzumab and Erlotinib as First-Line Therapy in Treating Women With Metastatic Breast Cancer Associated With HER2/Neu Overexpression
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-06-020; CDR0000069295; GENENTECH-OSI2365s; NCI-G02-2057
Record Dates: First submitted 2002-04-09; First posted 2003-01-27 (Estimated); Results first posted 2016-04-11 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2016-02

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- treatment (Experimental): please see intervention description
  Interventions: Biological: trastuzumab; Drug: erlotinib hydrochloride

INTERVENTIONS:
Biological: trastuzumab — Day 1 4mg/kg IV 2 mg/kg IV weekly.
  Other Names: Herceptin
Drug: erlotinib hydrochloride — 100 mg daily on Course 1 Day 2. After three weeks patients who have not experienced specific adverse events, dose will be escalated to 150 mg daily. Patients who have experienced specific adverse events dose will remain 100 mg daily or dose reduced as necessary per protocol.
  Other Names: OSI-774

SUMMARY:
RATIONALE: Monoclonal antibodies such as trastuzumab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Biological therapies such as erlotinib may interfere with the growth of tumor cells and slow the growth of the tumor. Combining trastuzumab with erlotinib may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining trastuzumab with erlotinib as first-line therapy in treating women who have metastatic breast cancer associated with HER2/neu overexpression.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and recommended phase II dose of erlotinib when combined with trastuzumab (Herceptin) as first-line therapy in women with metastatic breast cancer associated with HER2/neu overexpression. (Phase I closed to accrual as of 01/2004)
* Determine the safety profile of this regimen in these patients.
* Determine the rate and duration of objective response in patients treated with this regimen.
* Determine the pharmacologic behavior of this regimen in these patients.
* Determine time to disease progression and duration of survival in patients treated with this regimen.
* Correlate the antitumor activity of this regimen with epidermal growth factor receptor expression in these patients.

OUTLINE: This is a dose-escalation study of erlotinib. (Phase I closed to accrual as of 01/2004).

Patients receive oral erlotinib once daily beginning on day 2 and trastuzumab (Herceptin) IV over 30-90 minutes (1-4 hours after erlotinib) once weekly beginning on day 1. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of erlotinib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, additional patients are treated at the recommended phase II dose.

Patients are followed every 2 months.

PROJECTED ACCRUAL: A total of 3-18 patients will be accrued for the phase I portion (closed to accrual as of 01/2004) and 27-81 patients will be accrued for the phase II portion of this study.

ELIGIBILITY:
Inclusion Criteria:

* Women aged > 18 years
* Histologically documents metastatic breast cancer
* HER2 positive using Fluorescence In Situ Hybridization (FISH)
* For phase I, patients who have previously received treatment for their metastatic disease are allowed to participate.
* For the phase II portion of the study, patients must have measureable disease (> 2 cm; > 1 cm on spiral CT scan)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* A life expectancy of > 3 months
* Use of effective means of contraception

Exclusion Criteria:

* For Phase II, prior cytotoxic chemotherapy and/or prior Herceptin for their metastatic disease. Prior treatment in the adjuvant setting is allowed.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2001-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Britten, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States

REFERENCES:
- [Result] Britten CD, Finn RS, Bosserman LD, Wong SG, Press MF, Malik M, Lum BL, Slamon DJ. A phase I/II trial of trastuzumab plus erlotinib in metastatic HER2-positive breast cancer: a dual ErbB targeted approach. Clin Breast Cancer. 2009 Feb;9(1):16-22. doi: 10.3816/CBC.2009.n.003. PMID 19299235

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Phase 1; Treatment Phase 2: trastuzumab: Day 1 4mg/kg IV 2 mg/kg IV weekly.
  erlotinib hydrochloride: 100 mg daily on Course 1 Day 2. After three weeks patients who have not experienced specific adverse events, dose will be escalated to 150 mg daily. Patients who have experienced specific adverse events dose will remain 100 mg daily or dose reduced as necessary per protocol.
Period: Overall Study
Arm/Group | Treatment Phase 1 | Treatment Phase 2
Started | 16 | 11
Completed | 15 | 7
Not Completed | 1 | 4
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 0 | 3

BASELINE CHARACTERISTICS:
Population: enrolled subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Phase 1 | Treatment Phase 2 | Total
Number analyzed (Participants) | 16 | 11 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 9 | 23
  >=65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 11 | 27
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 11 | 7 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 16 | 11 | 27

OUTCOME MEASURES:

1. Primary Outcome: The Objective Response Rate as Defined as Stable Disease or the Rate of Complete and Partial Responses Determined on Two Consecutive Occasions Greater Than or Equal to 4 Weeks Apart.
Description: Complete Response:
  The disappearance of all signs of cancer in response to treatment. This does not always mean the cancer has been cured. Also called complete remission.
  Partial Response:
  A decrease in the size of a tumor, or in the extent of cancer in the body, in response to treatment. Also called partial remission.
Time Frame: 5 years
Population: 12 patients with measurable disease and no prior trastuzumab in the metastatic setting considered evaluable at the recommended phase II dose level. 2 from phase 1 and 10 from phase 2 Excluded : 14 from Phase I: no measureable disease or previous trastuzumab. Phase II: Withdrawn due to disease complications
Measure: Number; unit: participants
Groups:
- Treatment Phase 1 Plus Phase 2: trastuzumab: Day 1 4mg/kg IV 2 mg/kg IV weekly.
  erlotinib hydrochloride: 150 mg daily.
Arm/Group | Treatment Phase 1 Plus Phase 2
Number analyzed (Participants) | 12
participants
  Partial Response | 4
  Stable Disease | 1

2. Secondary Outcome: Duration of Objective Response
Time Frame: 5 years
Population: Subjects that achieved objective response (4). All were from phase II.
Measure: Number; unit: participants
Arm/Group | Treatment Phase 1 Plus Phase 2
Number analyzed (Participants) | 4
participants
  greater than 6 months | 4
  greater than 2 years | 2

3. Secondary Outcome: Incidence of Adverse Events
Time Frame: 5 years
Population: subjects evaluated for Serious Adverse Events (SAEs)
Measure: Number; unit: participants affected by SAEs
Groups:
- Treatment Phase 1 Plus Phase 2: trastuzumab: Day 1 4mg/kg IV 2 mg/kg IV weekly.
  erlotinib hydrochloride: 50mg daily, 100 mg daily and 150 mg daily.
Arm/Group | Treatment Phase 1 Plus Phase 2
Number analyzed (Participants) | 27
participants affected by SAEs | 16

4. Secondary Outcome: Serum Concentration of Herceptin at Specified Time-points.
Time Frame: 4 months
Measure: Mean (95% Confidence Interval); unit: mcg/mL
Groups:
- Treatment Phase 2: trastuzumab: Day 1 4mg/kg IV 2 mg/kg IV weekly.
  erlotinib hydrochloride:150 mg daily.
Arm/Group | Treatment Phase 2
Number analyzed (Participants) | 10
mcg/mL
  Day 7 peak | 98.4 [64.8 to 132]
  Day 7 trough | 46 [32.2 to 59.8]
  Day 14 peak | 86 [67.4 to 105]
  Day 14 trough | 46.9 [31.4 to 62.4]
  Day 21 peak | 88.3 [66.9 to 110]
  Day 21 trough | 50.8 [35.6 to 66]

5. Primary Outcome: Recommended Dose for Phase II
Time Frame: treatment period
Population: patients who have not experienced specific adverse events, dose will be escalated to 150 mg daily. Patients who have experienced specific adverse events dose will remain 100 mg daily or dose reduced as necessary per protocol.
Measure: Number; unit: participants receiving each dose
Arm/Group | Treatment Phase 1
Number analyzed (Participants) | 14
participants receiving each dose
  50 dose mg/day | 6
  100 dose mg/day | 3
  150 dose mg/day | 5

ADVERSE EVENTS:
Time Frame: 9.4 years
Arm/Group | Treatment Phase 1 Plus Phase 2
Serious Adverse Events (participants affected / at risk) | 16/27
Other Adverse Events (participants affected / at risk) | 22/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Phase 1 Plus Phase 2 (N=27)
dehydration/pain management (Gastrointestinal disorders) | 1 (1)
Dyspnea (Cardiac disorders) | 6 (6)
hypertension with headache (Cardiac disorders) | 1 (1)
pain/chest pressure/SOB (Cardiac disorders) | 1 (1) — back pain/neck pain/chest pressure-palpitations/shortness of breath
LVEF less than the lower limit of normal (Cardiac disorders) | 2 (2)
progressive brain mets (General disorders) | 2 (2)
gastroenteritis (Gastrointestinal disorders) | 1 (1) — gastroenteritis (per co-investigator, due to food poisoning)
maculopapular rash (Skin and subcutaneous tissue disorders) | 1 (1)
subendocardial myocardial infarction (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Phase 1 Plus Phase 2 (N=27)
alopecia (Skin and subcutaneous tissue disorders) | 4 (4)
anemia (Blood and lymphatic system disorders) | 3 (3)
anorexia (Gastrointestinal disorders) | 12 (12)
diarrhea (Gastrointestinal disorders) | 22 (22)
dry skin (Skin and subcutaneous tissue disorders) | 10 (10)
dysgeusia (Gastrointestinal disorders) | 4 (4)
dyspepsia (Gastrointestinal disorders) | 3 (3)
elevated transaminases (Metabolism and nutrition disorders) | 3 (3)
epistaxis (Blood and lymphatic system disorders) | 3 (3)
fatigue (General disorders) | 11 (11)
fever (General disorders) | 3 (3)
headache (General disorders) | 4 (4)
nausea (Gastrointestinal disorders) | 10 (10)
pruitus (Skin and subcutaneous tissue disorders) | 13 (13)
stomatitis (Gastrointestinal disorders) | 10 (10)
rash (Skin and subcutaneous tissue disorders) | 22 (22)
vomiting (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No